CLINICAL TRIAL: NCT05183139
Title: An Open-Label, Non-Comparative, Two-Cohort, Multicenter Study to Evaluate the Effectiveness and Safety of Ixazomib (NINLARO®) in Combination With Pomalidomide and Dexamethasone (IPd, Cohort A) or With Lenalidomide and Dexamethasone (IRd, Cohort B) in Patients With Relapsed/Refractory Multiple Myeloma Previously Receiving a Parenteral Proteasome Inhibitor-based Treatment Regimen (US MM-7)
Brief Title: A Multicenter In-class Transition Study of Ixazomib Combined With Pomalidomide and Dexamethasone or With Lenalidomide and Dexamethasone in Adults With Relapsed/Refractory Multiple Myeloma
Acronym: US MM-7
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision (no enrollment)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C16063
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; pomalidomide; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Ixazomib 4 mg + Pomalidomide 4 mg + Dexamethasone 40 mg (Experimental): Ixazomib 4 mg (3 mg for participants with moderate or severe hepatic impairment, severe renal impairment, or end-stage renal disease requiring dialysis), capsules, orally, on Days 1, 8, and 15, along with pomalidomide 4 mg, capsules, orally from Days 1 to 21 and dexamethasone 40 mg (20 mg if the participant is over 75 years of age), tablets, orally on Days 1, 8, 15, and 22 of each 28-day cycle, for a maximum of 39 cycles or until disease progression or unacceptable toxicity leading to discontinuation of ixazomib or to a change in regimen. Participants who were taking modified doses of pomalidomide or dexamethasone can start at that dose level in the study.
  Interventions: Drug: Ixazomib; Drug: Pomalidomide; Drug: Dexamethasone
- Cohort B: Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg (Experimental): Ixazomib 4 mg (3 mg for participants with moderate or severe hepatic impairment, severe renal impairment, or end-stage renal disease requiring dialysis), capsules, orally, on Days 1, 8, and 15, along with lenalidomide 25 mg capsules, orally, from Days 1 to 21 and dexamethasone 40 mg (20 mg if the participant is over 75 years of age), tablets, orally, on Days 1, 8, 15, and 22 of each 28-day cycle, for a maximum of 39 cycles or until disease progression or unacceptable toxicity leading to discontinuation of ixazomib or to a change in regimen. Participants who were taking modified doses of lenalidomide or dexamethasone can start at that dose level in the study.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
  Other Names: NINLARO
Drug: Pomalidomide — Pomalidomide capsules
  Other Names: POMALYST
  Arms: Cohort A: Ixazomib 4 mg + Pomalidomide 4 mg + Dexamethasone 40 mg
Drug: Lenalidomide — Lenalidomide capsules
  Other Names: REVLIMID
  Arms: Cohort B: Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Drug: Dexamethasone — Dexamethasone tablets

SUMMARY:
The main aim is to show that long-term use of ixazomib can improve symptoms of multiple myeloma and provide an effective long-term alternative treatment.

Participants will take ixazomib orally (by mouth) with pomalidomide and dexamethasone or lenalidomide and dexamethasone in 28-day treatment cycles. Participants will be treated for a maximum of 39 cycles but may continue to receive ixazomib beyond 39 cycles if they are benefiting from it. A follow-up study visit will occur 30 days after the last dose of ixazomib. Participants will be monitored for up to 3 years.

DETAILED DESCRIPTION:
The main objective is to determine whether an in-class transition (iCT) from a parenteral proteasome inhibitor (PI) regimen to an all-oral ixazomib(NINLARO) regimen can improve outcomes and provide an effective long-term alternative treatment for participants with relapsed and/or refractory multiple myeloma.

The drug being tested in this study is called ixazomib (NINLARO). Ixazomib is being tested to treat people who have relapsed and/or refractory multiple myeloma (R/R MM). This study will look at the efficacy and safety of ixazomib in participants with R/R MM who were previously receiving parenteral proteasome inhibitor (PI)-based therapy in combination with pomalidomide or with lenalidomide, and who undergo in-class transition to an oral ixazomib-based combination containing either pomalidomide (cohort A) or lenalidomide (cohort B).

The study will enroll approximately 140 patients. Participants will be enrolled to one of the two treatment groups, depending on whether they are transitioning from a pomalidomide- or lenalidomide- based regimen:

* Cohort A: Ixazomib 4 mg + Pomalidomide 4 mg + Dexamethasone 40 mg
* Cohort B: Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg

Participants who are >75 years of age at time of enrollment will be instructed to take 20 mg dexamethasone. For participants with moderate or severe hepatic impairment, severe renal impairment, or end-stage renal disease requiring dialysis, the recommended starting dose of ixazomib is 3 mg which can be further reduced to 2.3 mg at investigator's discretion.

This multi-center trial will be conducted at approximately 30 study centers across the United States. The overall duration of this study is approximately 5 years or until all participants have died, have been lost to follow-up, or completion of the study by the sponsor, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

1. Has a diagnosis of multiple myeloma (MM) using current IMWG diagnostic criteria, and are relapsed or refractory to 1 to 3 prior lines of therapy*.

   a. Has completed 3 or 4 cycles of a parenteral proteasome inhibitor (PI), and lenalidomide- or pomalidomide-based regimen and achieved a response of ≥ partial response (PR) with no evidence of disease progression as defined by IMWG criteria. This lead-in therapy to in-class transition (iCT) is not included as part of the 1 to 3 prior lines and should be completed no more than 28 days prior to initiation of IRd or IPd in this study.

   Those with light chain myeloma and free light chain (FLC) only may be enrolled if they previously met or currently meet the criteria for a diagnosis of MM.

   *A line of therapy is defined as one or more cycles of a planned treatment program. This may consist of one or more planned cycles of single-agent therapy or combination therapy, as well as a sequence of treatments administered in a planned manner. For example, a planned treatment approach of induction therapy followed by autologous stem-cell transplantation, followed by maintenance is considered one line of therapy. Autologous and allogenic transplants are permitted.
2. Has a diagnosis of non-secretory disease as long as the participant has a marker of disease that can be followed serially and assessed for response.
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status of 0, 1, or 2 at the time of enrollment.

Exclusion criteria

1. Has Grade >2 peripheral neuropathy (PN), or Grade 2 PN with pain on clinical examination.
2. Has not adequately recovered from other non-neuropathy AEs related to prior therapy in the opinion of the investigator at the time of enrollment.
3. Is pomalidomide refractory.
4. Has primary light chain amyloidosis (AL). Those with MM and concurrent AL are allowed.
5. Has known central nervous system involvement by MM.
6. Has infection requiring systemic antibiotic therapy or other serious infection within 14 days before enrollment.
7. Has ongoing or active systemic infection, active hepatitis B or C virus infection, or known positive status for human immunodeficiency virus.
8. Has been diagnosed or treated for another malignancy within 2 years before enrollment or has previously been diagnosed with another malignancy and has any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
9. Has previously been treated with ixazomib or participated in a study with ixazomib whether treated with ixazomib or not.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 5 years
  PFS is defined as the time from the date of the first administration of the study drug regimen ixazomib with pomalidomide and dexamethasone or ixazomib with lenalidomide and dexamethasone (IPd/IRd) to the date of the first documentation of disease progression before the start of next line of therapy based on local laboratory results and the investigator's assessment using modified International Myeloma Working Group (IMWG) response criteria or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Percentage of Participants Maintaining or Achieving PR, Very Good Partial Response (VGPR), or Complete Response (CR) | Up to approximately 5 years
  Percentage of participants with PR, VGPR, and CR will be determined based on local laboratory results and investigator's assessment using modified IMWG response criteria. CR: No immunofixation on serum/urine, disappearance of soft tissue plasmacytomas, <5% plasma cells in bone marrow. Participants with measurable disease only by serum free light chain (SFLC) level, normal FLC ratio of 0.26 to 1.65 in addition to CR criteria required. VGPR: Serum/urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% decrease in serum M-protein with urine M-protein <100 milligram per 24 hours (mg/24 hrs). If disease measurable only by SFLC, ≥90% decrease in difference between involved and uninvolved free light chain (dFLC) levels in addition to VGPR criteria required. PR: ≥50% reduction of serum M-protein and ≥90% reduction in urine M-protein or to <200 mg/24 hrs, or a ≥50% decrease in dFLC. If present at Baseline, ≥50% reduction in size of soft tissue plasmacytomas required.
Time to Progression (TTP) | Up to approximately 5 years
  TTP is defined as the time from the date of the first administration of the study drug regimen (IPd/IRd) to the date of the first documentation of disease progression based on local laboratory results and the investigator's assessment using modified IMWG response criteria.
Duration of Therapy (DoT 1) | Up to approximately 5 years
  DoT 1 is defined as the date of the first administration of the parenteral PI-based regimen to the date of the last administration of any of the three drugs in the study drug regimen.
Duration of Therapy (DoT 2) | Up to approximately 5 years
  DoT 2 is defined as the time from the date of the first administration of the study drug regimen (IPd or IRd) to the date of the last administration of any of the three drugs in the study drug regimen.
Duration of PI Therapy | Up to approximately 5 years
  Duration of parenteral PI therapy is defined as the time from the date of the first administration of the parenteral PI therapy of the regimen preceding the study drug regimen (IPd or IRd) to the date of the last administration of ixazomib therapy
Duration of Ixazomib Therapy | Up to approximately 5 years
  Duration of ixazomib therapy is defined as the time from the date of the first administration of ixazomib to the date of the last administration of ixazomib therapy.
Relative Dose Intensity (RDI) for Each Drug in the Treatment Regimen | Up to approximately 5 years
  RDI for each drug in the study drug regimen (IPd/IRd) is defined as 100 × (Total amount of dose taken)/(Total prescribed dose of treated cycles), where total prescribed dose equals (dose prescribed at enrollment) × number of prescribed doses per cycle × the number of treated cycles.
Percentage of Participants who Experience at Least One Treatment Emergent Adverse Event (TEAE) | Up to approximately 5 years
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/